CLINICAL TRIAL: NCT06831266
Title: Comparison of the Effects of High-Intensity Interval Exercise Training and Moderate-Intensity Continuous Exercise Training in Prediabetic Individuals: Single-Blind Randomized Controlled Study
Brief Title: Effects of Exercise Prediabetic Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ahsen Şenol, Lecturer, University of Kyrenia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETK00-2023-0184
Record Dates: First submitted 2025-01-29; First posted 2025-02-18 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Prediabetes / Type 2 Diabetes
Keywords: exercise; anti-inflammatory markers; aerobic capacity
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Masking Description: Masked for biomarker evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT High Intensity Interval Training (Experimental): High-intensity interval training (HIIT) is a type of training that involves repeated bouts of high intensity effort interspersed by recovery times.
  Interventions: Other: High Intensity Interval Training (HIIT)
- MICT Moderate Intensity Continuous Training (Active Comparator): Moderate Intensity Continuous Training (MICT) consists of performing aerobic exercise at a constant and moderate intensity for a prolonged duration.
  Interventions: Other: Moderate Intensity Continuous Training (MICT)

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) — 1 minute interval, 1 minute active recovery
  5 minutes warm-up - 3 minutes cool-down will be done at 60% of peak heart rate.
  Weeks 1-2: Loading at an intensity of 85% of peak heart rate, active recovery at an intensity of 60% of peak heart rate 4x1
  Weeks 2-7: Loading at an intensity of 90% of peak heart rate, active recovery at an intensity of 60% of peak heart rate 6x1
  Weeks 8-12: Loading at an intensity of 90% of peak heart rate, active recovery at an intensity of 60% of peak heart rate 8x1
  Other Names: High Intensity Interval Training
  Arms: HIIT High Intensity Interval Training
Other: Moderate Intensity Continuous Training (MICT) — 5 minutes warm-up - 3 minutes cool-down will be done at 60% of peak heart rate.
  Weeks 1-2: Loading at 65% of peak heart rate intensity (22 minute)
  Weeks 2-7: Loading at 75% of peak heart rate intensity (30 minute)
  Weeks 8-12: Loading at 75% of peak heart rate intensity (38 minute)
  Other Names: Moderate Intensity Continuous Training
  Arms: MICT Moderate Intensity Continuous Training

SUMMARY:
The aim of this study was to determine the effects of two different exercise protocols on body composition, aerobic capacity, blood lipid profile, some biomarkers, quality of life and exercise beliefs in participants at risk of diabetes.

DETAILED DESCRIPTION:
After being informed about the study and possible risks, all participants who gave written informed consent and met the eligibility requirements will be randomly assigned to 2 separate groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-60 years old
* HbA1c value between 5.7%-6.4%
* BMI>24,9 kg/m²
* Being sedentary
* Not on any diet

Exclusion Criteria:

* Insulin and derivative drug use
* Uncontrolled hypertension
* History of heart disease
* History of MI or stroke

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
HbAc | 12 weeks
  It is the amount of glycosylated hemoglobin in the blood.

SECONDARY OUTCOMES:
HDL | 12 weeks
  It is the amount of high-density lipoprotein in the blood.
LDL level LDL | 12 weeks
  It is the amount of low-density lipoprotein in the blood.
CRP | 12 weeks
  C-reactive protein is a protein produced in the liver.
Total cholesterol | 12 weeks
  Cholesterol is a lipid that is necessary for the construction of cell membranes in the body and the production of some hormones and vitamin D.
Triglyceride | 12 weeks
  It is a type of fat molecule found in the bloodstream and is used as the body's energy source.
Irisin | 12 weeks
  Irisin, defined as a myokine, is the proteolytic product of fibronectin type III domain 5 protein.
Adiponectin | 12 weeks
  Adiponectin is a protein hormone and adipokine, which is involved in regulating glucose levels and fatty acid breakdown.
IL-6 | 12 weeks
  Interleukin-6 is an endogenous chemical involved in inflammation and B cell maturation.
Resistin | 12 weeks
  Resistin is a hormone secreted from fat cells.
Kemerin | 12 weeks
  It is a protein that is involved in many metabolic events such as adipogenesis, angiogenesis and glucose homeostasis, including the chemoattractant function of the belt.
Osteocalcin | 12 weeks
  Osteocalcin is a bone-specific protein found in osteoblasts.
Leptin | 12 weeks
  Leptin is a hormone that acts on the hypothalamus through negative feedback secreted from fat cells, suppressing food intake and increasing energy expenditure.
TNF-alpha | 12 weeks
  Tumor necrosis factor alpha is a chemical messenger produced by the immune system that initiates inflammation.
Cardiometabolic risk level | 12 weeks
  Cardiometabolic risk has been defined as a cluster of metabolic and cardiovascular abnormalities, including abdominal obesity, insulin resistance, hypertension, dyslipidemia, and atherosclerosis, that predispose individuals to cardiovascular disease and type 2 diabetes.
Body composition | 12 weeks
  Body composition describes the amount of fat, bone, water and muscle in the body.
Aerobic capacity | 12 weeks
  Aerobic capacity is the capacity of large striated muscle groups to adapt to work using energy obtained from aerobic metabolism.
Exercise Health Belief Model Scale | 12 weeks
  Exercise Health Belief Model Scale is a 5-point Likert-type scale consists of 32 items.The scale consists of 5 factors and there is no reverse item. The highest and lowest score on the scale is 160 and 32, respectively. Higher scores indicate higher level of exercise health belief.
Short Form-36 Questionnaire | 12 weeks
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. SF-36 measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. High scores indicate good health status.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap Malkoç, Study Director — Eastern Mediterranean University
Locations (2):
- Turkey (Türkiye) (2):
  - University of Kyrenia Hospital, Mersin, Kyrenia
  - Eastern Mediterranean University, Mersin

IPD SHARING:
Plan to Share IPD: No